CLINICAL TRIAL: NCT04306393
Title: Nitric Oxide Gas Inhalation Therapy for Mechanically Ventilated Patients With Severe Acute Respiratory Syndrome Caused by SARS-CoV2: a Randomized Clinical Trial.
Brief Title: Nitric Oxide Gas Inhalation in Severe Acute Respiratory Syndrome in COVID-19
Acronym: NOSARSCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Xijing Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Niguarda Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Medical Doctor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO-SARS-COVID-19
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: SARS (Severe Acute Respiratory Syndrome); Coronavirus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient is blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Inhaled Nitric Oxide until PaO2/FiO2 >/= 300 mmHg
  Interventions: Drug: Nitric Oxide Gas
- Control Group (No Intervention)

INTERVENTIONS:
Drug: Nitric Oxide Gas — 80 ppm of inhaled nitric oxide for 48 hours, followed by 40 ppm, followed by weaning before stop.
  Weaning criteria: maintenance of a PaO2/FiO2 ratio >/= 300 for at least 24 hours consecutively.
  Arms: Treatment Group

SUMMARY:
Severe acute respiratory syndrome (SARS-CoV2) due to novel Coronavirus (2019-nCoV) related infection (COVID-19) is characterized by severe ventilation perfusion mismatch leading to refractory hypoxemia. To date, there is no specific treatment available for 2019-nCoV. Nitric oxide is a selective pulmonary vasodilator gas used in as a rescue therapy in refractory hypoxemia due to acute respiratory distress syndrome (ARDS). In-vitro and clinical evidence indicate that inhaled nitric oxide gas (iNO) has also antiviral activity against other strains of coronavirus. The primary aim of this study is to determine whether inhaled NO improves oxygenation in patients with hypoxic SARS-CoV2. This is a multicenter single-blinded randomized controlled trial with 1:1 individual allocation

DETAILED DESCRIPTION:
Severe acute respiratory syndrome (SARS-CoV-2) due to novel Coronavirus (2019-nCoV) related infection (COVID-19) is characterized by severe ventilation perfusion mismatch leading to refractory hypoxemia. To date, there is no specific treatment available for 2019-nCoV. Nitric oxide is a selective pulmonary vasodilator gas used as a rescue therapy in refractory hypoxemia due to acute respiratory distress syndrome (ARDS). In has also shown in-vitro and clinical evidence that inhaled nitric oxide gas (iNO) has antiviral activity against other strains of coronavirus.

The primary aim of this study is to determine whether inhaled NO improves oxygenation in patients with hypoxic SARS-CoV2.

This is a multicenter randomized controlled trial with 1:1 individual allocation. Patients will be blinded to the treatment.

Intubated patients admitted to the intensive care unit with confirmed SARS-CoV-2 infection and severe hypoxemia will be randomized to receive inhalation of NO (treatment group) or not (control group). Treatment will be stopped when patients are free from hypoxemia for more than 24 hours.

ELIGIBILITY:
Inclusion criteria: (1) Adult patients, >/= 18 year-old; (2) Patients admitted to the ICU; (3) Patients who are intubated and mechanically ventilated; (4) Confirmed diagnosis of SARS-CoV2 by positive rt-PCR.

Exclusion criteria: (1) Patients intubated for more than 72 hours from initiation of the treatment gas; (2) Subjects enrolled in another interventional research study; (3) Physician of record opposed to enrolling the patient due to perceived safety concerns; or any condition that does not allow the protocol to be followed safely; (4) Subjects with past medical history of lung malignancy or pneumonectomy or lung transplant; (5) Subjects receiving a tidal volume < 3 cc/kg of ideal body weight at the time of enrollment; (6) Subjects with severe burns involving more than 40% of Total Body Surface Area; (7) Subjects that have experienced cardiac arrest with CPR for longer than 30 minutes; (8) Subjects with a presumed severe deficit in cerebral function with fixed dilated pupil; (9) Subjects receiving renal replacement therapy at the time of enrollment; (10) Subjects who have an impaired ability to ventilate without assistance; (11) Subjects who have a history of malignancy or other irreversible disease/conditions with a 6-month mortality > 50%; (12) Subjects not fully committed to full support at the time of enrollment; (13) Subject receiving inhaled nitric oxide gas prior to enrollment; (14) Subject's hospital admission unrelated to COVID-19.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Change of arterial oxygenation at 48 hours from enrollment | 48 hours
  Difference within groups in terms of PaO2/FiO2 ratio. If a patient dies during the first 48 hours of treatment, the last available blood gas analysis will be used.

SECONDARY OUTCOMES:
Time to reach normoxemia during the first 28 days after enrollment | 28 days
  Time to recover gas exchange to a PaO2/FiO2 =/> 300 for at least 24 hours during the first 28 days after enrollment, within each group and comparison between groups. If the patient dies before day 28, the patient will be considered as "never recovered".
Proportion of SARS-nCoV-2 free patients during the first 28 days after enrollment | 28 days
  Daily proportion of patients with a PaO2/FiO2 ratio > 300 for at least 24 hours within each group and comparison between groups. If a patient dies before day 28, the patient will be considered as "never recovered".
Survival at 28 days from enrollment | 28 days
  Proportion of patients surviving at 28 days within each group and comparison between groups.
Survival at 90 days from enrollment | 90 days
  Proportion of patients surviving at 90 days within each group and comparison between groups.

OTHER OUTCOMES:
Daily oxygenation in the two groups until day 28 | 28 days
  Expressed as PaO2/FiO2 ratio within each group and comparison between groups.
Need for new renal replacement therapy during the first 28 days | 28 days
  Proportion of patients needing RRT within each group and comparison between groups.
Mechanical support of circulation during the first 28 days | 28 days
  Proportion of patients needing mechanical support of circulation (i.e., ECMO, intra-aortic balloon pump, VADs) within each group and comparison between groups.
Days free of vasopressors during the first 28 days | 28 days
  Average days without need for vasopressors within each group and comparison between groups.
Ventilator-free days at 28 days | 28 days
  Average days without need for mechanical ventilation within each group and comparison between groups.
Time to SARS-CoV-2 rt-PCR negative in upper respiratory tract specimen | 28 days
  Time to obtain first negative upper respiratory tract sample in the 2019-nCoV rt-PCR assay. Average within groups and comparison between groups.
ICU-free days at 28 days | 28 days
  Average days out of ICU within each group and comparison between groups.
ICU length of stay | 90 days
  Average days of ICU admission within each group and comparison between groups.
SARS-CoV-2 Viral Load in Sputum | 28 days
  Number of copies of SARS-CoV-2 Viral Load measured with rt-PCR on sputum samples within each group and comparison between groups.
SARS-CoV-2 Viral Load in Plasma | 28 days
  Number of copies of SARS-CoV-2 Viral Load measured with rt-PCR on blood samples within each group and comparison between groups.
Acute Kidney Injury at 28 days | 28 days
  Proportion of patients with acute kidney injury and severity of acute kidney injury within each group and comparison between groups.
Daily Vasoactive Inotropic Score | 28 days
  Daily calculation of the vasoactive inotropic score in each group and comparison between groups.
Requirement for VV-ECMO | 28 days
  Proportion of patients requiring venous-venous extracorporeal membrane oxygenation within each group and comparison between groups.
Daily Sequential Organ Failure Assessment | 28 days
  Daily calculation of the sequential organ failure assessment within each group and comparison between groups.
Hospital-free days at 28 days | 28 days
  Average days after hospital discharge within each group and comparison between groups.
Hospital length of stay | 90 days
  Average days of hospital stay within each group and comparison between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Study Director — Massachusetts General Hospital
Locations (5):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - Louisiana State University Health Shreveport, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
- Danderyd Sjukhus AB, Danderyd, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gibson LE, Fenza RD, Lang M, Capriles MI, Li MD, Kalpathy-Cramer J, Little BP, Arora P, Mueller AL, Ichinose F, Bittner EA, Berra L, G Chang M. Right Ventricular Strain Is Common in Intubated COVID-19 Patients and Does Not Reflect Severity of Respiratory Illness. J Intensive Care Med. 2021 Aug;36(8):900-909. doi: 10.1177/08850666211006335. Epub 2021 Mar 30. PMID 33783269
- [Derived] Lei C, Su B, Dong H, Bellavia A, Fenza RD, Fakhr BS, Gianni S, Grassi LG, Kacmarek R, Morais CCA, Pinciroli R, Vassena E, Berra L. Protocol of a randomized controlled trial testing inhaled Nitric Oxide in mechanically ventilated patients with severe acute respiratory syndrome in COVID-19 (SARS-CoV-2). medRxiv [Preprint]. 2020 May 24:2020.03.09.20033530. doi: 10.1101/2020.03.09.20033530. PMID 32511534